CLINICAL TRIAL: NCT04438421
Title: Efficacy of a Filming Formulation of Hydrogen Peroxide and Hyaluronic Acid (BMG0703) in the Treatment of Inflammation and Bleeding Caused by Gingivitis, Compared to Placebo and 0.2% Chlorhexidine. A Randomised Controlled Clinical Trial.
Brief Title: Efficacy of Hyaluronic-acid and Hydrogen-Peroxide Mouthwash in Gingivitis Treatment
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Chiara Occhipinti, Professor, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BMG0703_ORC_May 2019 v.0
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Gingivitis; Bleeding Gum
Keywords: Gingivitis; Bleeding; Plaque; Tartar
MeSH Terms: conditions — Gingivitis; Gingival Hemorrhage; Hemorrhage; Plaque, Amyloid; Dental Calculus | interventions — Hydrogen Peroxide; Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: 50 subjects affected with gingivitis, caused by accumulation of plaque and/or tartar, will be selected and enrolled in this study. Subsequently, subjects will be equally divided and randomly allocated to either the test group or the control group.
Who Masked: Participant, Investigator
Masking Description: The products will be packaged in such a way that they are not recognizable neither by the operator, nor by the patient. Each package will be assigned a number that in turn will refer to the type of the product. The association between the number and type of the product will be collected by another operator according to the association carried out by a dedicated software. The operator who will deliver the product will be informed about the type only at the end of the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BMG0703 (Experimental): Subjects will then be given the test product, BMG0703, to be used twice a day after meals and after normal oral hygiene procedures. Next, the subjects will be re-evaluated after 3 days and after one month.
  Interventions: Drug: Filming mouthwash formulation, enriched with Hydrogen Peroxide and Hyaluronic Acid
- Chlorhexidine 0.2% (Active Comparator): Subjects will then be given a 0.2% Chlorhexidine product, to be used twice a day after meals and after normal oral hygiene procedures. Next, the subjects will be reevaluated after 3 days and after one month.
  Interventions: Drug: Chlorhexidine mouthwash
- Placebo Product (Placebo Comparator): Subjects will then be given a placebo product, to be used twice a day after meals and after normal oral hygiene procedures. Next, the subjects will be reevaluated after 3 days and after one month.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Filming mouthwash formulation, enriched with Hydrogen Peroxide and Hyaluronic Acid — Subjects will then be given the test product, BMG0703, to be used twice a day after meals and after normal oral hygiene procedures. Next, the subjects will be re-evaluated after 3 days and after one month.
  Other Names: BMG0703
  Arms: BMG0703
Drug: Chlorhexidine mouthwash — Subjects will then be given Chlorhexidine 0.2%mouthwash, as an active comparator, to be used twice a day after meals and after normal oral hygiene procedures. Next, the subjects will be re-evaluated after 3 days and after one month.
  Other Names: Chlorhexidine 0.2%
  Arms: Chlorhexidine 0.2%
Drug: Placebo — Subjects will then be given a placebo product to be used twice a day after meals and after normal oral hygiene procedures. Next, the subjects will be re-evaluated after 3 days and after one month.
  Other Names: Placebo product
  Arms: Placebo Product

SUMMARY:
A clinical study to evaluate the efficacy and safety of a mouthwash containing Hydrogen Peroxide, Sodium Hyaluronate and Glycine in the prevention and management of complications associated gingivitis by film forming action.

DETAILED DESCRIPTION:
50 subjects will be enrolled, who show with gingivitis caused by accumulation of plaque and/or tartar selected consecutively. Subsequently, subjects will be equally divided and randomized into the test group or control group.

During the three examinations, the subjects will undergo the collection of bleeding and plaque indices according to Silness J & Loe H 3,4. Four surfaces per tooth (vestibular, lingual/palatal, mesial, distal) will be considered.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 12 and 50 years
* Presence of gingivitis caused by accumulation of plaque/tartar
* Acceptance of informed consent

Exclusion Criteria:

* subjects suffering from HIV
* subjects suffering from hepatitis
* serious systemic diseases preventing the use of specific dental therapies
* acute and/or chronic infectious diseases
* inability to provide consent
* use of topical or systemic drugs
* inability to follow post-intervention hygiene instructions
* smokers

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Change in Bleeding index | 0, 3, 30 days
  Subjects will undergo the measurement of bleeding index according to Silness J & Loe. Four surfaces per tooth (vestibular, lingual/palatal, mesial, distal) will be considered.
  Data will be collected based on four possible clinical conditions:
  Code 0: absence of bleeding during probing depth measurement; Code 1: absence of bleeding during probing depth measurement, presence of redness and oedema; Code 2: presence of bleeding during probing depth measurement with redness and oedema; Code 3: spontaneous bleeding
  Higher score means worse outcome.
Change in Plaque index | 0, 3, 30 days
  Subjects will undergo the measurement of plaque index according to Silness J & Loe. Four surfaces per tooth (vestibular, lingual/palatal, mesial, distal) will be considered.
  Data will be collected based on four possible clinical conditions:
  Code 0: absence of plaque; Code 1: presence of plaque not visible to the naked eye but evidenced by the periodontal probe passage; Code 2: presence of plaque at the level of the gingival margin; Code 3: abundant presence of plaque at the level of the gingival margin and/or the rest of the dental surface.
  The sum of the values of the four surfaces examined, divided by the very number of surfaces, will give the plaque and bleeding index value for each individual tooth. The sum of the indices of each examined tooth divided by the total number of teeth examined will indicate the overall plaque and bleeding index of the subject at that time.

CONTACTS AND LOCATIONS:
Overall Officials: Giampietro Farronato, Professor, Principal Investigator — University of Milan; Gianguido Cossellu, Fellow, Principal Investigator — University of Milan
Locations (1):
- UOC Maxillofacial Surgery and Odontology, University of Milan, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Protocol data available in PDF format upon request

REFERENCES:
- [Background] Axelsson P, Nystrom B, Lindhe J. The long-term effect of a plaque control program on tooth mortality, caries and periodontal disease in adults. Results after 30 years of maintenance. J Clin Periodontol. 2004 Sep;31(9):749-57. doi: 10.1111/j.1600-051X.2004.00563.x. PMID 15312097
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464
- [Background] Loe H. The Gingival Index, the Plaque Index and the Retention Index Systems. J Periodontol. 1967 Nov-Dec;38(6):Suppl:610-6. doi: 10.1902/jop.1967.38.6.610. No abstract available. PMID 5237684
- [Background] Marchetti E, Tecco S, Caterini E, Casalena F, Quinzi V, Mattei A, Marzo G. Alcohol-free essential oils containing mouthrinse efficacy on three-day supragingival plaque regrowth: a randomized crossover clinical trial. Trials. 2017 Mar 31;18(1):154. doi: 10.1186/s13063-017-1901-z. PMID 28359280
- [Background] van der Weijden F, Slot DE. Oral hygiene in the prevention of periodontal diseases: the evidence. Periodontol 2000. 2011 Feb;55(1):104-23. doi: 10.1111/j.1600-0757.2009.00337.x. No abstract available. PMID 21134231